CLINICAL TRIAL: NCT00002930
Title: Whole-Body 18F-Fluorodeoxyglucose Positron Emission Tomography to Measure the Response to Induction Chemotherapy of Potentially Resectable Lung and Esophageal Carcinomas
Brief Title: PET Scan in Patients With Lung and Esophageal Cancers That May Be Removed by Surgery
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Diagnostic
Other Study IDs: 96-079; P30CA008748 (NIH); MSKCC-96079; NCI-G97-1334
Record Dates: First submitted 1999-11-01; First posted 2004-03-12 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Esophageal Cancer; Lung Cancer
Keywords: stage I non-small cell lung cancer; stage II non-small cell lung cancer; stage I esophageal cancer; stage II esophageal cancer; stage III esophageal cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer
MeSH Terms: conditions — Esophageal Neoplasms; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Magnetic Resonance Spectroscopy; Fluorodeoxyglucose F18

INTERVENTIONS:
Procedure: positron emission tomography
Radiation: fludeoxyglucose F 18

SUMMARY:
RATIONALE: Imaging procedures, such as fludeoxyglucose F 18 positron emission tomography (PET) scans, may improve the ability to detect lung and esophageal cancer or their recurrence.

PURPOSE: Phase II/III trial to study the effectiveness of fludeoxyglucose F 18 PET scans in measuring response to induction chemotherapy in patients with esophageal and lung cancer that may be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine whether whole body fludeoxyglucose F 18 (F-18 2-fluoro-2-deoxy-D-glucose; FDG) positron emission tomography (PET) can quantitate the response to induction (preoperative) chemotherapy in patients with esophageal or non-small cell lung cancer (NSCLC) by correlating changes in PET scan images with surgical staging, frequency of complete resection, disease-free survival, and overall survival. II. Correlate PET scan results with the multiple conventional complementary imaging modalities of thoracic and/or abdominal CT, bone scans, and cranial MRI. III. Evaluate the use of PET scanning to uncover disease sites undetected by current imaging modalities.

OUTLINE: This is a nonrandomized study. The choice of chemotherapeutic regimen is at the discretion of the medical oncologist. If the tumor is resectable after treatment with chemotherapy, the patients undergoes the appropriate resection as defined by the thoracic surgeon. All patients have positron emission tomography (PET) scans done within 2 weeks before the first dose of chemotherapy and again about 2-3 weeks after the third or fourth dose of chemotherapy. Patients are asked to not eat or drink 6 hours before coming into the hospital for the PET scan. They are administered an injection of a solution of fluorodeoxyglucose F 18 (FDG) and then undergo a PET scan.

PROJECTED ACCRUAL: An estimated 75 patients (50 lung cancer and 25 esophageal cancer patients) will be accrued into this protocol over 24-30 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed esophageal or non-small cell lung carcinoma Esophageal cancer: Biopsy proven esophageal carcinoma considered acceptable for curative esophageal resection Lung cancer: Stages IA-IIIB, T(any)N(any)M0 disease without pleural effusion, which constitutes locally advanced lung cancer Must be candidates for induction chemotherapy followed by surgical resection

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 70-100% Life expectancy: Not specified Hematopoietic: WBC at least 4,000/mm3 Platelet count at least 160,000/mm3 Hepatic: Bilirubin no greater than 1.0 mg/dL Renal: Creatinine no greater than 1.5 mg/dL Creatinine clearance greater than 65 mL/min Other: Not pregnant Adequate contraception required of all fertile female patients

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: No prior surgical mediastinal staging such as prior mediastinoscopy or Chamberlain procedures See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 1996-12; Primary Completion 2002-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J. Downey, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States